CLINICAL TRIAL: NCT00758485
Title: A Randomized, Safety-assessor Blinded Trial Comparing 4.0 mg.Kg-1 Sugammadex With Placebo in Adult Subjects Scheduled for Surgery Requiring Profound Neuromuscular Blockade
Brief Title: Comparing 4.0 mg.Kg-1 Sugammadex With Placebo in the Reversal of Profound Neuromuscular Blockade (P05767)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05767; 2008-002518-23 (EudraCT Number); 19.4.316 (Other: Organon Protocol ID); MK-8616-004 (Other: Merck Protocol ID)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia; Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugammadex (Experimental): Participants receiving 4.0 mg.kg-1 Sugammadex at a target depth of NMB of 1-2 PTC after the last dose of rocuronium
  Interventions: Drug: Sugammadex
- Placebo (Placebo Comparator): Participants receiving Placebo (0.9% NaCl) at a target depth of NMB of 1-2 PTC after the last dose of rocuronium
  Interventions: Drug: 0.9% sodium chloride (NaCl)

INTERVENTIONS:
Drug: Sugammadex — At a target depth of NMB of 1-2 PTC after the last dose of rocuronium, a bolus dose of 4.0 mg.kg-1 sugammadex (volume based on the actual body weight of the participant) will be administered, within 10 seconds into a fast running venous infusion.
  Other Names: Org 25969; SCH 900616; MK-8616; Bridion®
  Arms: sugammadex
Drug: 0.9% sodium chloride (NaCl) — At a target depth of NMB of 1-2 PTC after the last dose of rocuronium, a bolus dose of placebo (0.9% NaCl, volume based on the actual body weight of the participant) will be administered, within 10 seconds into a fast running venous infusion.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The current trial was designed to demonstrate faster recovery in participants undergoing elective surgeries requiring profound neuromuscular blockade induced by rocuronium to a fourth twitch/first twitch (T4/T1) ratio of 0.9, after reversal of a target depth of neuromuscular blockade (NMB) of 1-2 Post Tetanic Count (PTC) by 4.0 mg.kg-1 Sugammadex compared to Placebo, to evaluate the safety of 4.0 mg.kg-1 Sugammadex and to evaluate the Operating Room (OR) and Post Anesthetic Care Unit (PACU) length of stay for these participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants
* American Society of Anesthesiologists (ASA) class 1, 2 or 3
* Age >=18 years
* Scheduled to undergo a surgery requiring profound NMB such as cardiovascular, gynaecologic, neurologic and thoracic surgical procedures under general anesthesia requiring neuromuscular relaxation with rocuronium for endotracheal intubation and if applicable maintenance of NMB in a position allowing neuromuscular monitoring
* Given written informed consent

Exclusion Criteria:

* Participants known or suspected to have neuromuscular disorders affecting NMB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

REFERENCES:
- [Result] Rahe-Meyer N, Berger C, Wittmann M, Solomon C, Abels EA, Rietbergen H, Reuter DA. Recovery from prolonged deep rocuronium-induced neuromuscular blockade: A randomized comparison of sugammadex reversal with spontaneous recovery. Anaesthesist. 2015 Jul;64(7):506-12. doi: 10.1007/s00101-015-0048-0. Epub 2015 Jul 1. PMID 26126940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 sites in Germany from November 2008 to May 2009.
Groups:
- Sugammadex: Participants receiving 4.0 mg.kg-1 Sugammadex at a target depth of neuromuscular blockade (NMB) of 1-2 Post Tetanic Count (PTC) after the last dose of rocuronium
- Placebo: Participants receiving Placebo (0.9% sodium chloride[NaCl]) at a target depth of NMB of 1-2 PTC after the last dose of rocuronium
Period: Overall Study
Arm/Group | Sugammadex | Placebo
Started | 70 | 70
TREATED | 69 | 68
Completed | 69 | 67
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not Treated | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Placebo | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (17) | 57 (14) | 57 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 48 | 43 | 91

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Investigational Medicinal Product (IMP, Sugammadex or Placebo) to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (a percentage that is expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB), with a higher ratio indicating a greater recovery from NMB. In this study, twitch responses were recorded until the T4/T1 Ratio reached >=0.9, the minimum acceptable ratio that indicated complete recovery from NMB. A shorter time to recovery of the T4/T1 Ratio >=0.9 indicates a faster recovery from NMB.
Time Frame: From Start of IMP Administration to Recovery of the T4/T1 Ratio to 0.9 (estimated from ~2 minutes up to ~90 minutes)
Population: The Intent-to-Treat (ITT) Population consisted of all participants who received either Sugammadex or Placebo and had at least one efficacy measurement. Imputed recovery times were used in cases of missing times.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Groups:
- Sugammadex: Participants receiving 4.0 mg/kg-1 Sugammadex at a target depth of NMB of 1-2 Post Tetanic Count (PTC) after the last dose of rocuronium
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 69 | 65
minutes | 2.2 [1.9 to 2.5] | 89.8 [80.1 to 100.7]

2. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (a percentage that is expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating a greater recovery from NMB.
Time Frame: From Start of IMP Administration to Recovery of the T4/T1 Ratio to 0.7 (estimated from ~1 minute up to ~70 minutes)
Population: The ITT Population consisted of all participants who received either Sugammadex or Placebo and had at least one efficacy measurement. Imputed recovery times were used in cases of missing times.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 69 | 65
minutes | 1.6 [1.4 to 1.8] | 70.1 [62.7 to 78.4]

3. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.8
Description: as for outcome 2
Time Frame: From Start of IMP Administration to Recovery of the T4/T1 Ratio to 0.8 (estimated from ~2 minutes up to ~80 minutes)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 69 | 65
minutes | 1.8 [1.6 to 2.0] | 78.8 [70.2 to 88.5]

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of IMP
Description: The All Subjects Treated Population consisted of all randomized participants who received IMP.
Arm/Group | Sugammadex | Placebo
Serious Adverse Events (participants affected / at risk) | 4/69 | 4/68
Other Adverse Events (participants affected / at risk) | 44/69 | 48/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=69) | Placebo (N=68)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=69) | Placebo (N=68)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4)
Flatulence (Gastrointestinal disorders) | 4 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (9) | 11 (12)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Procedural Nausea (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 29 (30) | 32 (33)
Wound Complication (Injury, poisoning and procedural complications) | 11 (13) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 7 (7) | 5 (5)
Sleep Disorder (Psychiatric disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No